CLINICAL TRIAL: NCT05253339
Title: A Single-center Randomized Controlled Trial Comparing the Standard Method and Target-controlled Infusion as a Method of Administering Cefoxitin, Which is Used to Prevent Surgical Site Infections in Colorectal Surgical Patients
Brief Title: The Expected Advantage of Administering Prophylactic Antibiotics Using Target- Concentration Controlled Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Seoul Business Agency (Unknown)
Responsible Party: Principal Investigator, Byung-Moon Choi, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0180
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Anti-bacterial Agents; Pharmacokinetics; General Surgery

STUDY DESIGN:
Intervention Model Description: When administering cefoxitin, the standard administration method and the target concentration control injection method are randomly assigned 1:1.
Who Masked: Participant
Masking Description: Only the patient is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard administration method (Active Comparator): Drug: Cefoxitin, Device: not applicable (standard method)
  Two grams of cefoxitin (JW Pharmaceutical Co., Ltd., Seoul, South Korea) was dissolved in 50 mL of normal saline and administered for about 10 min before skin incision.
  Interventions: Procedure: Standard administration method
- Target controlled infusion (TCI) (Experimental): Drug: Cefoxitin, Device: TCI Syringe pump
  Two grams of cefoxitin were dissolved in 50 mL of normal saline to give a concentration of 40 mg/mL. Before skin incision, cefoxitin was infused with a TCI syringe pump (Pilot Anesthesia 2, Fresenius vial, France), which was connected to a personal computer by an RS232c cable and controlled with TCI software (Asan pump, version 2.1.3; Bionet Co. Ltd., Seoul, Korea, http://www.fit4nm.org/download, last accessed: 27 August, 2012). Target concentrations of total concentrations were set to 80 μg/mL.
  Interventions: Procedure: target-controlled infusion (one of the administration methods)

INTERVENTIONS:
Procedure: target-controlled infusion (one of the administration methods) — a method of administering cefoxitin while maintaining a constant target concentration.
  Arms: Target controlled infusion (TCI)
Procedure: Standard administration method — Standard method of administering cefoxitin in the current clinical setting
  Arms: Standard administration method

SUMMARY:
Preoperative antimicrobial prophylaxis is a key element for the prevention of surgical site infection, the most common type of nosocomial infection in surgical patients. Prophylactic antibiotics are selected depending on the type of surgery, and first- or second-generation cephalosporins have been mainly used. Cefoxitin, a second-generation cephalosporin with anaerobic activity, has been used in various clinical settings as a prophylactic antibiotic for colorectal surgery. Cefoxitin is generally dissolved in normal saline and intravenously administered for a short time of 5-10 minutes before skin incision. However, there are several drawbacks to the current dosing strategy. First, the dose of cefazolin is determined by a "rule of thumb", and there is controversy over whether 1 g or 2 g is appropriate, with the opinion that 2 g being more appropriate prevailing. Second, the standard administration method unnecessarily induces a concentration higher than the concentration required to prevent surgical site infection. Third, significant covariates that can affect the maintenance of MIC during surgery are not considered. The target-concentration controlled infusion (TCI) method can be a viable alternative administration method for antibiotics. The TCI method enables individual customized administration according to the covariates (i.e., weight, creatinine clearance) included in the pharmacokinetic parameters; also, although with some variability, the drug can be administered while maintaining the target concentration. The aim of this study was to evaluate the effectiveness of administering cefoxitin in patients undergoing colorectal surgery with a syringe pump equipped with a target concentration control injection function

DETAILED DESCRIPTION:
Parenteral antimicrobial prophylaxis before abdominal surgery for preventing surgical site infection (SSI) is a well-established clinical practice. Prophylactic antibiotics are selected depending on the type of surgery, and first- or second-generation cephalosporins have been mainly used. These antibiotics are generally dissolved in normal saline and intravenously administered for a short time of 5-10 min before skin incision. However, the conventional administration strategy has several problems. First, the dose of antibiotics does not take into account the patients' physical characteristics such as body weight, age, and renal function. Considering that the dosages of practically all drugs used in clinical fields are determined based on body weight, it may be necessary to improve the dosing strategy to reflect the patient's physical characteristics based on the effectiveness and safety of the antibiotic. Second, the plasma concentration of cephalosporin becomes excessively high at the end of the administration, which is more pronounced in patients with low body weight. The minimal inhibitory concentrations (MIC) for each antibiotic are well-characterized; however, a pilot simulation study showed that at the end of the administration, the plasma concentration of cefazolin was 20 times higher than its MIC. It is difficult to exclude the possibility that concentrations higher than necessary may cause harm to patients. Third, the bactericidal activity of an antibiotic is apparent when its free plasma concentration is maintained above the MIC. Using the conventional administration method, there is a period during the entire surgical period in which the concentration decreases below the MIC unless redosing is performed. Taken together, it is necessary to develop a method for administering a prophylactic antibiotic to overcome these problems.

The target-controlled infusion (TCI) is a method of administering a drug while maintaining a target concentration and has been used for more than 20 years for administering hypnotic agents and opioids during general anesthesia. Because the infusion rate is continuously recalculated by an infusion algorithm mounted on the TCI infusion pump to maintain the target concentration, the infusion rate is not fixed and changes over time. The patient's specific characteristics such as body weight and creatinine clearance can be included in the pharmacokinetic parameters so that even when administered for the same duration and the same target concentration, the actual dosage varies for each patient and allows for personalized administration. Thus, the population pharmacokinetic parameters of a drug are required to administer the drug by the TCI method.

The risk of SSI varies depending on the type of surgery, and colorectal surgery is regarded as having a high risk of SSI because of the possibility of wound contamination from bowel contents. Accordingly, the incidence of SSI has been reported to be 4-10% in colon surgery and 3-27% in rectal surgery. In the case of colorectal surgery, the optimal prophylactic antibiotic has not been unified into one agent. Cefoxitin, a second-generation cephalosporin with anaerobic activity, has been used in various clinical settings as a prophylactic antibiotic for colorectal surgery.

The aim of this study was to evaluate the effectiveness of administering cefoxitin in patients undergoing colorectal surgery with a syringe pump equipped with a target concentration control injection function

ELIGIBILITY:
Inclusion Criteria:

* over 20 years old
* Patients who are scheduled to undergo colon or rectal surgery
* Patients scheduled to receive cefoxitin as a prophylactic antibiotic

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to cefoxitin
* Patients with a history of receiving cefoxitin within 3 days of the scheduled surgery time
* Patients receiving therapeutic antibiotics
* eGFR < 30 ml/min/1.73m2

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2494 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
The incidence of surgical site infections | Within 30 days after the operation
  Surgical site infection (SSI) is an infection that occurs after surgery in the part of the body where the surgery took place. Superficial incisional SSI occurs just in the area of the skin where the incision was made. Deep incisional SSI occurs beneath the incision area in muscle and the tissues surrounding the muscles. Organ-space SSI includes infections involving any part of the anatomy that was opened or manipulated during an operation

SECONDARY OUTCOMES:
Total dose of cefoxitin | on the day of surgery
  Total amount of cefoxitin administered as prophylactic antibiotics. Redosing is performed every two hours after the first dose.

OTHER OUTCOMES:
The incidence of acute kidney injury | Within 7 days after the operation
  An increase in serum creatinine by ≥ 0.3 mg/dl within 48 h or an increase in serum creatinine to ≥ 1.5 times baseline within the previous 7 days or urine volume ≤ 0.5 ml/kg/h for 6 h

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Moon Choi, Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-Gu,, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HJ, Kim KM, Lee JL, Park IJ, Choi BM. A single-centre randomised controlled trial comparing the standard method and target-controlled infusion as a method of administering cefoxitin, which is used to prevent surgical site infections in colorectal surgical patients: study protocol. Trials. 2025 Jan 8;26(1):11. doi: 10.1186/s13063-025-08716-x. PMID 39780190